CLINICAL TRIAL: NCT03289949
Title: The Neurobiological Effect of 5-HT2AR Modulation
Acronym: NeuroPharm2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gitte Moos Knudsen (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Professor, DMsc, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: H-16026898
Record Dates: First submitted 2017-09-14; First posted 2017-09-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Basic Science
MeSH Terms: interventions — Psilocybin; Ketanserin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Project 1: Occupancy of psilocybin/ketanserin (Other): After baseline MRI & 5-HT2AR PET-imaging, participants will be allocated to undergo either one oral dose of psilocybine or one oral dose of ketanserin. After drug administration, participants will undergo two CIMBI-36 PET scans.
  Interventions: Drug: Psilocybine; Drug: Ketanserin
- Project 2: Long term effects of psilocybin (Other): After baseline MRI & CIMBI-36 PET-imaging, participants will receive one dose of oral psilocybine intervention. One and 12 weeks after dosing, participants will undergo post-intervention PET-scan.
  Subproject B: After baseline MRI & UCB-J PET-imaging, participants will receive one dose of oral psilocybine intervention. One week after dosing, participants will undergo post-intervention UCB-J PET-scan.
  Subproject C: After baseline MR imaging, participants will receive one dose of oral psilocybine (25 mg) or placebo. One month after dosing, participants will undergo a post-intervention MRI scan.
  Interventions: Drug: Psilocybine
- Project 3: Functional connectivity (Other): After baseline MRI scanning and CIMBI-36 PET, participants will undergo one psilocybine-intervention fMRI scan and one ketanserin-intervention fMRI scan. If P2 shows there are long term effects of psilocybine on 5-HT2AR levels, psilocybine will be fixed as the second intervention. If not, interventions will be randomized.
  Interventions: Drug: Psilocybine; Drug: Ketanserin

INTERVENTIONS:
Drug: Psilocybine — Oral dose of psilocybine.
  Other Names: Psilocybin
Drug: Ketanserin — Oral dose of ketanserin.
  Other Names: Ketensin
  Arms: Project 1: Occupancy of psilocybin/ketanserin; Project 3: Functional connectivity

SUMMARY:
The investigators wish to investigate neurobiological effects of serotonin 2A receptor modulation in healthy volunteers, contrasting effects of an agonist (psilocybin) and an antagonist (ketanserin). Magnetic resonance imaging (MRI) and positron emission tomography (PET) will be used as neuroimaging tools.

DETAILED DESCRIPTION:
This project applies an experimental medicine strategy coupled with human functional and molecular neuroimaging to elucidate the effects of 5-HT2A receptor (5-HT2AR) modulation on brain function and mood in healthy individuals. We compare psilocybin (5-HT2AR agonist) and ketanserin (5-HT2AR antagonist) effects on brain function to identify neural mechanisms mediating the clinical effects of psilocybin and, more broadly, to establish this comparative strategy as a pathway for delineating pharmacological effects on the brain in humans.

ELIGIBILITY:
Inclusion Criteria:

1) Healthy individuals above 18 years of age.

Exclusion Criteria (For Subprojects 1, 2a, 2b, and 3):

1. Presence of or previous primary psychiatric disease (DSM axis 1 or WHO ICD-10 diagnostic classifications) or in first-degree relatives.
2. Previous or present neurological condition/disease, significant somatic condition/disease or intake of drugs suspected to influence test results.
3. Non-fluent Danish language skills.
4. Vision or hearing impairment.
5. Previous or present learning disability.
6. Pregnancy.
7. Breastfeeding.
8. Contraindications in regard to MRI scanning.
9. Alcohol or drug abuse.
10. Allergy to test drugs.
11. Participation in studies in which participant has received more than 10 mSv of radiation or other significant exposure to radiation.
12. Abnormal ECG or intake of QT prolonging medication.
13. Previous significant side-effects in regard to hallucinogenic drugs.
14. Use of hallucinogenic drugs 6 months previous to inclusion.
15. Blood donation 3 months before and after project participation
16. Body weight under 50 kg.
17. Plasma ferritin levels outside normal range

Exclusion Criteria (For Subproject 2c):

1. Presence of or previous primary psychiatric disease (DSM IV axis 1 or WHO ICD-10 diagnostic classifications).
2. Presence of or previous primary psychiatric disease with psychosis symptoms or hypomania (DSM IV axis 1 [drug/alcohol abuse/dependence, schizophrenia and other psychoses] or WHO ICD-10 diagnostic classifications [F10-29, as well as F30-39 with psychotic symptoms, F60]) in first-degree relatives (parents or siblings).
3. Previous or present neurological condition/disease, significant somatic condition/disease or intake of drugs suspected to influence test results.
4. Non-fluent Danish language skills or pronounced vision or hearing impairment.
5. Previous or present learning disability.
6. Pregnancy.
7. Breastfeeding.
8. Contraindications in regard to MRI scanning.
9. Alcohol or drug abuse.
10. Allergy to test drugs.
11. Abnormal ECG or intake of QT prolonging medication.
12. Previous significant side-effects in regard to hallucinogenic drugs.
13. Previous use of hallucinogenic drugs.
14. Body weight under 45 kg.
15. Ethical concerns regarding the administration of a psychedelic drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Psilocin/ketanserin blood concentrations and 5-HT2A receptor occupancy (i.e., binding potential). | Change in Cimbi-36 binding potential from baseline PET to intervention PET 1 and PET 2 scans (same day for psilocybin, and two consecutive days for ketanserin).
  The investigators aim to model relations psilocin/ketanserin blood drug concentrations and receptor occupancy, using C11-Cimbi-36 PET imaging.
Effects of psilocybin on Cimbi-36 binding potential at baseline and at one and twelve weeks | Change in Cimbi-36 binding potential from baseline to one week post psilocybin (and potentially also at 12 weeks after psilocybin).
  Cimbi-36 PET scan binding potential at baseline and at one-week post psilocybin, and potentially also at 12 weeks post psilocybin.
Effects of psilocybin and ketanserin on brain function assessed with fMRI and PET | Changes in functional connectivity (fMRI) from Baseline MR to intervention MR scans for ketanserin (one or three weeks after baseline MR) and psilocybin (one or three weeks after baseline)
  Correlations between blood levels of ketanserin and psilocin and the estimated associated receptor occupancy with functional MRI neuroimaging data, including resting state networks. Changes in synaptic density will be assessed with 11C-UCB-J PET scans before and 1 week after psilocybin intervention.
Effects of psilocybin on UCB-J binding potential at baseline and at one week | Change in UCB-J binding potential from baseline to one week post psilocybin.
  Project 2, Subproject B. UCB-J PET scan binding potential at baseline and at one-week post psilocybin.
Effects of psilocybin on brain function assessed with fMRI at baseline and one month | Change in fMRI measures from baseline to one month post psilocybin
  Project 2, Subproject C. Resting-state and task-based fMRI measures at baseline and one month post psilocybin.
Anxiety Outcome Measure 1: Acute psychological effects as assessed using Challenging Experiences Questionnaire (CEQ). | Immediately post-intervention.
  Differences in CEQ scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Likert-scale ranging from 0 (Not all all) to 5 (Extremely; More than ever). Higher scores thus reflect a more challenging experience. Project 2, Subproject C. PsiloZonic.
Anxiety Outcome Measure 2: Acute psychological effects as assessed using 5D-Altered States of Consciousness (5D-ASC) scale. | Immediately post-intervention.
  Differences in 5D-ASC anxiety scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Visual analogue scale (VAS) scale ranging from 0 (No, not more than usually) to 100 (Yes, much more than usually). Higher scores on dimension anxiety thus reflect more anxiety. Project 2, Subproject C. PsiloZonic.
Anxiety Outcome Measure 3: Acute psychological effects as assessed using Extended Subjective Drug Intensity (eSDI) scale. | During intervention.
  Differences in eSDI anxiety scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Likert-scale ranging from 0 (Not all all) to 10 (Very much). Higher scores on item anxiety thus reflect more anxiety. Project 2, Subproject C. PsiloZonic.
Transformative Experiences Outcome Measure 1: Acute psychological effects as assessed using Mystical Type Experiences Questionnaire (MEQ) scale. | Immediately post-intervention.
  Differences in MEQ scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Likert-scale ranging from 0 (Not all all) to 5 (Extremely). Higher scores thus reflect a more profound mystical type experience. Project 2, Subproject C. PsiloZonic.
Transformative Experiences Outcome Measure 2: Acute psychological effects as assessed using Psychological Insights Questionnaire (PIQ) scale. | Immediately post-intervention.
  Differences in PIQ scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Likert-scale ranging from 0 (Not all all) to 5 (Extremely). Higher scores thus reflect more psychological insight. Project 2, Subproject C. PsiloZonic.
Transformative Experiences Outcome Measure 3: Acute psychological effects as assessed using Emotional Breakthrough Questionnaire (EBI) scale. | Immediately post-intervention.
  Differences in EBI scores between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Visual analogue scale (VAS) scale ranging from 0 (No, not more than usually) to 100 (Yes, much more than usually). Higher scores thus reflect more emotional breakthrough. Project 2, Subproject C. PsiloZonic.
Persisting Effects Outcome Measure 1: Persisting psychological effects as assessed using Persisting Effects Questionnaire (PEQ) scale. | One and three months post-intervention.
  Differences in PEQ scores will be assessed between groups (psilocybin with music compared to psilocybin without music). Effects are measured on a Likert-scale ranging from 0 (Not all all) to 5 (Extremely). Higher scores thus reflect more persisting effects. Project 2, Subproject C. PsiloZonic.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, Professor, Study Chair — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage) data will be available for neuroscience research community contingent on approval by scientific board.
Supporting Information: Study Protocol
Time Frame: Upon project completion
Access Criteria: All researchers can request access to data from the database by completing a standardized application form to provide detailed information about the specific database request. The application form and guidelines are available here. Please note that there are some formal requirements that must be fulfilled if the data request is from an international researcher. For example we do not have permission for sharing data outside of the EU, so researchers from a non-EU country will have to come here to work on the data instead.
URL: https://cimbi.dk/db